CLINICAL TRIAL: NCT00191061
Title: A Comparison of Duloxetine Dosing Strategies in The Treatment of Patients With Major Depression
Brief Title: A Comparison of Tolerability and Efficacy of Different Doses of Duloxetine for the Treatment of Major Depressive Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8950; F1D-US-HMDR
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2007-01-26 (Estimated); Status verified 2007-01

CONDITIONS: Depressive Disorder
MeSH Terms: conditions — Depressive Disorder | interventions — Duloxetine Hydrochloride

INTERVENTIONS:
Drug: duloxetine hydrochloride

SUMMARY:
The purpose of this study is to compare the tolerability and efficacy of different doses of duloxetine in patients with major depressive disorder.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients at least 18 years of age (male and/or female) who meet criteria for major depressive disorder (MDD) as defined by the Diagnostic and Statistical Manual for Mental Disorders Fourth Edition Text Revision (DSM-IV-TR). Patients may have comorbid Anxiety Disorders, except for Obsessive Compulsive Disorder
* Tests negative for pregnancy at the time of enrollment based on a serum pregnancy test and agrees to use a reliable method of birth control (for example, use of oral contraceptives or Norplant a reliable barrier method of birth control diaphragms with contraceptive jelly; cervical caps with contraceptive jelly; condoms with contraceptive foam; intrauterine devices; partner with vasectomy; or abstinence) during the study and for 1 month following the last dose of study drug.
* Hamilton Depression Rating 17 Item Scale (HAMD-17) greater than 15 at Visits 1 and 2.

Exclusion Criteria:

* Have any current Axis I disorder other than major depressive disorder (MDD), dysthymia, or any anxiety disorder; however, obsessive-compulsive disorder is excluded.
* Have any previous or current diagnosis of bipolar disorder, obsessive-compulsive disorder, schizophrenia, or other psychotic disorders.
* Lack of response of the current episode of major depression to two or more adequate courses of antidepressant therapy at clinically appropriate dose for a minimum of 4 weeks or, in the judgment of the investigator, the patient meets criteria for treatment-resistant depression.
* DSM-IV-TR-defined history of substance abuse or dependence within the past 6 months, excluding nicotine and caffeine.
* Patients judged to be at serious suicidal risk in the opinion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 640
Dates: Start 2004-10; Study Completion 2006-01

PRIMARY OUTCOMES:
The primary objective in the acute phase of this study is to compare the incidence of treatment-emergent nausea
for patients initially dosed at duloxetine 30 mg QD
(once-daily), versus duloxetine 60 mg QD.
The primary objective in the extension phase of this study is to compare efficacy in patients not meeting response criteria during the acute phase for patients dosed at duloxetine 60 mg QD versus duloxetine 120 mg QD.

SECONDARY OUTCOMES:
The secondary objective of greatest importance is to compare the incidence of treatment-emergent nausea
(as defined for the primary objective) for patients
initially dosed at duloxetine 30 mg QD, versus duloxetine 30 mg BID (twice-daily).
Additional secondary objectives include comparing the three initial dosing groups in regards to:Mean changes from baseline in the category total scores and individual items scores of the AMDP-5
The incidence and severity of adverse events using rates of spontaneously reported treatment-emergent adverse events, rates of discontinuations due to
adverse events, categorical changes in AMDP-5 items, mean changes and categorical changes in vital signs
as well as mean changes and rates of abnormal laboratory analytes
Mean changes from baseline in the HAMD17 total score, HAMD subscales, HAMD17 individual items, 30-item Inventory of Depressive Symptoms,
Clinician Rated (IDS-30) total score and individual items, Brief Pain Inventory items and interference
total score, Visual Analog Scales for pain, Clinical Global Impressions of Severity (CGI-Severity), Post-baseline means
on the Patient's Global Impression of Improvement (PGI-I), Remission rates (HAMD17 total score of less than 7),
and response rates (greater than 50% decrease from baseline on the HAMD17 total score).
- Sexual dysfunction, as measured by categorical changes (same, better, worse) and presence vs. absence, based on the patient global assessment of sexual functioning.
Time to onset of action in depression (30% improvement in Maier Subscale of HAMD) and painful physical symptoms (30% improvement in as measure by the BPI interference total score).

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (32):
- United States (32):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Little Rock, Arkansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Coral Springs, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jacksonville, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Miami, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Port Charlotte, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Boise, Idaho
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Edwardsville, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lafayette, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Terre Haute, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Metairie, Louisiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New Orleans, Louisiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Glen Burnie, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Belmont, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St Louis, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Clementon, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Princeton, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Albuquerque, New Mexico
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New York, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Olean, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Eugene, Oregon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Portland, Oregon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Philadelphia, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sioux Falls, South Dakota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Memphis, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Houston, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lake Jackson, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Charlottesville, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Midlothian, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Richmond, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seattle, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brown Deer, Wisconsin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., West Allis, Wisconsin

REFERENCES:
- [Derived] Perlis RH, Fijal B, Dharia S, Houston JP. Pharmacogenetic investigation of response to duloxetine treatment in generalized anxiety disorder. Pharmacogenomics J. 2013 Jun;13(3):280-5. doi: 10.1038/tpj.2011.62. Epub 2012 Jan 17. PMID 22249355
- [Derived] Kornstein SG, Dunner DL, Meyers AL, Whitmyer VG, Mallinckrodt CH, Wohlreich MM, Detke MJ, Hollandbeck MS, Greist JH. A randomized, double-blind study of increasing or maintaining duloxetine dose in patients without remission of major depressive disorder after initial duloxetine therapy. J Clin Psychiatry. 2008 Sep;69(9):1383-92. doi: 10.4088/jcp.v69n0905. PMID 19193339
- [Derived] Whitmyer VG, Dunner DL, Kornstein SG, Meyers AL, Mallinckrodt CH, Wohlreich MM, Gonzales JS, Greist JH. A comparison of initial duloxetine dosing strategies in patients with major depressive disorder. J Clin Psychiatry. 2007 Dec;68(12):1921-30. doi: 10.4088/jcp.v68n1213. PMID 18162024